CLINICAL TRIAL: NCT04976569
Title: Neuromodulation of Sleep Architecture by STN-DBS in Parkinsonian Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tsinghua University (Other)
Collaborators: Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Principal Investigator, Luming Li, : Director of National Engineering Laboratory for Neuromodulation, Tsinghua University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STN_DBS_Sleep_TsinghuaU
Record Dates: First submitted 2021-06-16; First posted 2021-07-26 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease; Sleep Disorder
MeSH Terms: conditions — Parkinson Disease; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBS Regulation Group (Experimental): All participants will receive STN-DBS sleep regulation.
  Interventions: Device: STN-DBS stimulation pattern change

INTERVENTIONS:
Device: STN-DBS stimulation pattern change — Deep brain stimulation (DBS) is an elective surgical procedure in which electrodes are implanted into certain brain areas.We use specific STN-DBS stimulation pattern to regulate sleep architecture.

SUMMARY:
Sleep disorder is one of the most burdensome non-motor symptoms in Parkinsonian patients. Typical manifestations include RBD, decreased sleep efficiency, decreased slow wave sleep, daytime sleepiness, increased sleep latency and wakefulness during sleep. Subthalamic nucleus (STN) deep brain stimulation (DBS) has been reported to improve sleep dysfunction in several studies, mostly due to its improvement in motor dysfunction. However, there are limited research about specific STN-DBS stimulation pattern for sleep architecture regulation, and whether suboptimal parameter combinations for motor has potential benefits for sleep improvement has not been studied. Here we use different parameter combination in STN-DBS, especially by changing stimulation contact and frequency, to explore the specific stimulation pattern for normalizing sleep architecture and increasing slow wave sleep.

DETAILED DESCRIPTION:
Investigators will enroll at least 5 subjects for this study. First, subjects will be clinically evaluated by motor, cognitive and sleep scales; Subsequently, the treatment window of each contact using unipolar stimulation will be tested both in high frequency (such as 130Hz) and low frequency (such as 80Hz), and the parameters of stimulation were determined under the premise of no obvious discomfort and optimal motor control. Different stimulation pattern (such as ventral contact stimulation) will be performed during the N2 phase combined with PSG and LFP recording during the patients' sleep, and switch to baseline stimulation pattern at the N3/N1/REM phase. Repeat these steps until the patient wake up naturally. Finally, the patients will be evaluated for motor function. Pre-surgery and post-surgery images will be used for reconstructing VTA of specific parameter combination. Functional MRI (fMRI) will be carried out to verify the connectivity change under optimal parameter combinations.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease: The diagnostic criteria for Parkinson's disease are the Clinical Diagnostic Criteria of UK PD Society Brain Bank Clinical Diagnostic Criteria or 2015 MDS Clinical Diagnostic Criteria for PD.All diagnoses of Parkinson's disease were made by three neurologists who were experienced in the field of movement disorders.
2. Bilateral STN-DBS has been implanted for more than 1 year, and stable drug therapy regimen and parameter program control regimen have been maintained for 6 weeks or more;
3. Patients with onset age of 50 years and above;
4. Do not use phenobarbital, chloral hydrate, benzodiazepines and non-benzodiazepines as sedatives and hypnotics at night.

Exclusion Criteria:

1. Patients who underwent pallidotomy and other brain surgery;
2. Other patients with secondary Parkinson's syndrome and Parkinsonism-plus syndrome;
3. Patients with other central nervous system and peripheral nervous system diseases;
4. Patients complicated with severe medical system diseases, patients with unstable vital signs and unable to tolerate clinical evaluation;
5. Patients with severe mental illness;
6. Use phenobarbital, chloral hydrate, benzodiazepines and non-benzodiazepines as sedatives and hypnotics at night;
7. Patients who cannot complete informed consent due to cognitive and communication barriers, or refuse to sign informed consent.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
ratio of slow wave sleep | through study completion, an average of 1 year
  The percentage of slow wave sleep
ratio of rem sleep | through study completion, an average of 1 year
  The percentage of rem sleep
Sleep Efficiency | through study completion, an average of 1 year
  The percentage of time a person sleeps, in relation to the amount of time a person spends in bed

SECONDARY OUTCOMES:
Motor Function Evaluation | through study completion, an average of 1 year
  Using MDS-UPDRS III to evaluation motor function both before and after whole night sleep to verify influence of different stimulation pattern on motor function during sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- National Engineering Laboratory for Neuromodulation, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No